CLINICAL TRIAL: NCT02713646
Title: Applied Research on Patients With Trigeminal Neuralgia by Multi-planar Reconstruction, Curved Planar Reconstruction and Magnetic Resonance Virtual Endoscopy
Brief Title: Magnetic Resonance Imaging Study on Patients With Trigeminal Neuralgia
Acronym: MRI-TN
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRF-2015-028
Record Dates: First submitted 2016-03-06; First posted 2016-03-21 (Estimated); Last update posted 2023-02-16 (Actual); Status verified 2020-02

CONDITIONS: Trigeminal Neuralgia
Keywords: MRI; Virtual Endoscopy; Pain Measurement
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- patients with primary trigeminal neuralgia
- healthy subjects

SUMMARY:
Up to now, multiplanar reconstruction (MPR) has been widely used to detect the neurovascular compressions (NVC) on the patients with idiopathic trigeminal neuralgia (ITN). However, due to lack of stereoscopic vision, this traditional method sometimes cannot meet the requirement on identifying the existence and details of NVC, especially when the aberrant vessels turn out to be delicate veins. The three-dimensional analytic techniques, such as curved planar reconstruction (CPR) and magnetic resonance virtual endoscopy (MRVE), may be helpful to improve the sensitivity and specificity on the demonstration of NVC with stereo and dynamic views, so as to assist to design the surgical plan.

Furthermore, the frequent finding of NVC on MRI studies of asymptomatic patients incited the creation of several strict criteria for the imaging diagnosis of NVC: the vessel must cross perpendicular to the long axis of the nerve, the nerve must be deviated or indented at the root entry zoon (REZ) by the vessel. Alternatively, morphological measurement of the nerve may correlate with the severity of facial pain due to atrophy of the nerve in most cases of ITN, and is likely secondary to the micro-structural abnormalities, such as axonal loss, demyelination, collagen deposition, etc. In this study, cross-sectional area (CSA) and volume (V) of the cisternal trigeminal nerve will be assessed to determine whether it can be a useful biomarker for predicting the degree of ITN.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis according to the International Classification of Headache Disorders criteria (3rd edition); 1 year disease duration at least.

Exclusion Criteria:

* Secondary causes of ITN; Precarious general health status; Percutaneous lesions or surgical treatments; Cardiac pacemaker or metal implants.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic trigeminal neuralgia patients prior to the surgery of microvascular decompression (MVD) or Gamma Knife radiofrequency ablation (GKRFA)
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline V (mm3) at 12 months | 0, 12 months
  Baseline V (mm3) refers to the volume of the cisternal trigeminal nerve prior to the surgical treatment. Meanwhile, the study endpoint is 12 months after the operation, which need another measurement of V.
  Measurements of V will be performed using Medical Image Processing, Analysis, and Visualization software (MIPAV, http://mipav.cit.nih.gov/). The measurements start from the point where the nerves enter the pons to an imaginary demarcation made at the entrance of the nerves into Meckel's cave. The trigeminal nerves are manually delineated in each traverse section. The V will be automatically calculated with the MIPAV software.
Change from Baseline CSA (mm2) at 12 months | 0, 12 months
  Baseline CSA (mm2) refers to the cross sectional area of the cisternal trigeminal nerve prior to the surgical treatment. Meanwhile, the study endpoint is 12 months after the operation, which need another measurement of CSA. The CSA is calculated at 5 mm from the entry of the trigeminal nerve into the pons in an image plane perfectly perpendicular to the course of each nerve, which also need using a mouse-driven cursor in MIPAV software.

SECONDARY OUTCOMES:
Sensitivity and Specificity of Detection of Neurovascular Compression by MPR Compared with Surgical Findings | 0 (baseline)
  Severity of neurovascular compression, which will be judged by MPR, is defined as follows: 1 = no compression; 2 = contact by a vessel; 3 = indentation by a vessel; and 4 = nerve displacement or distortion by a vessel, and the results of MPR need to be compared with the intraoperative findings to obtain the sensitivity and specificity, respectively.
Sensitivity and Specificity of Detection of Neurovascular Compression by CPR Compared with Surgical Findings | 0 (baseline)
  Severity of neurovascular compression, which will be judged by CPR, is the same criterion as that in the Outcome 3, and the results of CPR need to be compared with the intraoperative findings to obtain the sensitivity and specificity, respectively.
Sensitivity and Specificity of Detection of Neurovascular Compression by MRVE Compared with Surgical Findings | 0 (baseline)
  Severity of neurovascular compression, which will be judged by MRVE, is the same criterion as that in the Outcome 3, and the results of MRVE need to be compared with the intraoperative findings to obtain the sensitivity and specificity, respectively.
Change from Baseline Visual Analog Score (VAS) for Pain at 12 months | 0, 12 months
  Baseline VAS will be evaluated by Visual Analog Scale for Pain prior to the operations. Graphic formats for the VAS can be obtained online: http:// www.amda.com/tools/library/whitepapers/hospiceinltc/appendix-a.pdf. Meanwhile, the study endpoint is 12 months after the operation, which need another measurement of VAS.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhang, M.D. & Ph.D., Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- 3.0-T MRI scanner (Signa HDxt; GE Medical Systems, WI, USA), Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Leal PR, Barbier C, Hermier M, Souza MA, Cristino-Filho G, Sindou M. Atrophic changes in the trigeminal nerves of patients with trigeminal neuralgia due to neurovascular compression and their association with the severity of compression and clinical outcomes. J Neurosurg. 2014 Jun;120(6):1484-95. doi: 10.3171/2014.2.JNS131288. Epub 2014 Apr 18. PMID 24745706
- [Result] Erbay SH, Bhadelia RA, O'Callaghan M, Gupta P, Riesenburger R, Krackov W, Polak JF. Nerve atrophy in severe trigeminal neuralgia: noninvasive confirmation at MR imaging--initial experience. Radiology. 2006 Feb;238(2):689-92. doi: 10.1148/radiol.2382042214. PMID 16436823
- [Result] Borges A, Casselman J. Imaging the trigeminal nerve. Eur J Radiol. 2010 May;74(2):323-40. doi: 10.1016/j.ejrad.2010.02.006. Epub 2010 Mar 12. PMID 20227216
- [Result] Satoh T, Omi M, Nabeshima M, Onoda K, Date I. Severity analysis of neurovascular contact in patients with trigeminal neuralgia: assessment with the inner view of the 3D MR cisternogram and angiogram fusion imaging. AJNR Am J Neuroradiol. 2009 Mar;30(3):603-7. doi: 10.3174/ajnr.A1409. Epub 2008 Nov 27. PMID 19039051
- [Derived] Xu H, Jia L, Wang Y, Han W, Li D, Zhang M, Wang Y. Abnormalities of cortical morphology and structural covariance network in the patients with primary trigeminal neuralgia: a preliminary clinical study. Neurol Sci. 2025 Sep;46(9):4527-4535. doi: 10.1007/s10072-025-08360-y. Epub 2025 Jul 15. PMID 40663271
- [Derived] Xu H, Liu Y, Zeng WT, Fan YX, Wang Y. Distinctive cortical morphological patterns in primary trigeminal neuralgia: a cross-sectional clinical study. Neuroradiology. 2024 Feb;66(2):207-216. doi: 10.1007/s00234-023-03257-z. Epub 2023 Nov 25. PMID 38001310
- [Derived] Wang Y, Yang Q, Cao D, Seminowicz D, Remeniuk B, Gao L, Zhang M. Correlation between nerve atrophy, brain grey matter volume and pain severity in patients with primary trigeminal neuralgia. Cephalalgia. 2019 Apr;39(4):515-525. doi: 10.1177/0333102418793643. Epub 2018 Aug 7. PMID 30086682